CLINICAL TRIAL: NCT04333979
Title: Effect of Drain Usage on Patient Comfort on Laparoscopic Sleeve Gastrectomy
Brief Title: The Effect of Drain Use on Patient Comfort in Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ersin Gündoğan, Doctor- lecturer-Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-181
Record Dates: First submitted 2019-01-08; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Obesity, Morbid
Keywords: obesity; VAS; Pain; Laparoscopy; Sleeve
MeSH Terms: conditions — Obesity, Morbid; Obesity; Pain | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain replacement (Experimental): Effects of drainage
  Interventions: Other: Drainage
- Drain not placed (No Intervention): Effects of not using drain

INTERVENTIONS:
Other: Drainage — Using drain after operation
  Arms: Drain replacement

SUMMARY:
Introduction Laparoscopic sleeve gastrectomy surgeon; Have become increasingly morbid obesity treatment methods with improvements in minimally invasive surgery. Ensuring patient comfort and early return to life are the criteria that should be given priority in this treatment method. The purpose of this study is to determine the use of drain, which closely affects these criteria; And the effect on patient comfort.

DETAILED DESCRIPTION:
Question the necessity of routine use of drain in Laparoscopic sleeve gastrectomy surgeon

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese patients

Exclusion Criteria:

* - Cirrhotic patients, those under 18 years of age, additional intraabdominal surgeries during Laparoscopic sleeve gastrectomy and those who had previously undergone obesity surgery (revision surgery) were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Pain Intensity measure | 6 months
  self reported pain intensity morning. item is scored 0-10 ( 0: no pain- 10: pain as bad as can be)

IPD SHARING:
Plan to Share IPD: No